CLINICAL TRIAL: NCT05188729
Title: A Phase 2, Multicenter, Open-label, Proof-of-concept Study With Safety Run-in to Evaluate the Safety, Pharmacokinetics, and Efficacy of VP-315 in Adult Subjects With Basal Cell Carcinoma
Brief Title: Open-Label Proof of Concept Study of VP-315 in Basal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verrica Pharmaceuticals Inc. (Industry)
Collaborators: Instat Clinical Research (Unknown); HeartcoR Solutions (Unknown); Myonex (Unknown); Vial Health Technology, Inc (Unknown); OncoBay Clinical (Unknown); Q2 Solutions (Industry); Canfield Scientific (Unknown); Veristat (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VP-315-201
Record Dates: First submitted 2021-12-13; First posted 2022-01-12 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Basal Cell Carcinoma; Skin Cancer; Cancer of the Skin, Basal Cell; Cancer of the Skin; Carcinoma
Keywords: Skin Cancer; BCC; Neoplasm; Epithelial
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms; Carcinoma; Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicenter, dose-escalating study. Eligible subjects will be enrolled sequentially.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1 - Cohort 1: Dose Escalation VP-315 2 mg (Experimental): Cohort 1: Starting total daily dose of VP-315 will be 2 mg. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 2 mg on Day 1, 3 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
  Interventions: Drug: Part 1: VP-315 3 Day Dosing/Week
- Part 1 - Cohort 2: Dose Escalation VP-315 3 mg (Experimental): Cohort 2: Starting total daily dose of VP-315 will be 3 mg. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 3 mg on Day 1, 4 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
  Interventions: Drug: Part 1: VP-315 3 Day Dosing/Week
- Part 1 - Cohort 3: Dose Escalation VP-315 4 mg (Experimental): Cohort 3: Starting total daily dose of VP-315 will be 4 mg. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 4 mg on Day 1, 5 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
  Interventions: Drug: Part 1: VP-315 3 Day Dosing/Week
- Part 1 - Cohort 4: Dose Escalation VP-315 5 mg (Experimental): Cohort 4: Starting total daily dose of VP-315 will be 5 mg. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 5 mg on Day 1, 6 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
  Interventions: Drug: Part 1: VP-315 3 Day Dosing/Week
- Part 1 - Cohort 5: Dose Escalation VP-315 6 mg (Experimental): Cohort 5: Starting total daily dose of VP-315 will be 6 mg. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 6 mg on Day 1, 7 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
  Interventions: Drug: Part 1: VP-315 3 Day Dosing/Week
- Part 1 - Cohort 6: Dose Escalation VP-315 7 mg (Experimental): Cohort 6: Starting total daily dose of VP-315 will be 7 mg. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 7 mg on Day 1, 8 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
  Interventions: Drug: Part 1: VP-315 3 Day Dosing/Week
- Part 1 - Cohort 7: Dose Escalation VP-315 8 mg (Experimental): Cohort 7: Starting total daily dose of VP-315 will be 8 mg. Subjects will receive once daily doses of 8 mg for up to 3 days in a 7-day treatment week (e.g., 8 mg on Day 1, 8 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
  Interventions: Drug: Part 1: VP-315 3 Day Dosing/Week
- Part 2 - Cohort 1: Optimal Dosing Regimen of 3 daily doses of VP-315, 4 mg loading dose (Experimental): VP-315 once-daily dosing of 8 mg with a loading dose of half the target dose of 8 mg (i.e. 4 mg) only on W1D1; all remaining doses will be the full target dose without a loading dose. Subjects will be treated until the lesion is necrosed, for a maximum of 2 weeks (W1D1, W1D2, W1D3 and W2D1, W2D2, W2D3 - up to 6 total doses).
  Interventions: Drug: Part 2: VP-315 3 Day Dosing/Week - Loading Dose
- Part 2 - Cohort 2: Optimal Dosing Regimen of 3 daily doses of VP-315 no loading dose (Experimental): VP-315 once-daily dosing of 8 mg on all treatment days (i.e., NO LOADING dose on W1D1) for up to 3 consecutive daily doses/week until the lesion is necrosed, for a maximum of 2 weeks (W1D1, W1D2, W1D3 and W2D1, W2D2, W2D3 - up to 6 total doses).
  Interventions: Drug: Part 2: VP-315 3 Day Dosing/Week - No Loading Dose
- Part 2 - Cohort 4: Optimal Dosing Regimen of 2 daily doses of VP-315 8 mg (split dose) (Experimental): VP-315 once-daily dosing of 8 mg, administered on 2 consecutive days in one week (W1D1, W1D2). The planned dosing regimen will be a split dose of VP-315 for all treatments. The 500μL (8 mg) dose will be divided into 2 injections given at least 15 minutes and no more than 30 minutes apart, with 30% (150 μL) administered in the first injection and the remaining 70% (350 μL) with the second injection. Treatment for a second Target Lesion may begin on D1 of the next week (W2D1, W2D2). Each individual target lesion is treated for the assigned 2 days only (regardless of necrosis status). Up to 2 target lesions may be treated - up to 4 total doses.
  Interventions: Drug: Part 2: VP-315 2 Day Dosing/Week - Split Dose
- Part 2 - Cohort 5: Optimal Dosing Regimen of 3 daily doses of VP-315 8 mg (split dose) (Experimental): VP-315 once-daily dosing of 8 mg, administered on 3 consecutive days in one week (W1D1, W1D2, W1D3). The planned dosing regimen will be a split dose of VP-315 for all treatments. The 500μL (8 mg) dose will be divided into 2 injections given at least 15 minutes and no more than 30 minutes apart, with 30% (150 μL) administered in the first injection and the remaining 70% (350 μL) with the second injection. Treatment for a second target lesion may begin on D1 of the next week (W2D1, W2D2, W2D3). Each individual target lesion is treated for the assigned 3 days only (regardless of necrosis status). Up to 2 target lesions may be treated - up to 6 total doses.
  Interventions: Drug: Part 2: VP-315 3 Day Dosing/Week - Split Dose

INTERVENTIONS:
Drug: Part 1: VP-315 3 Day Dosing/Week — 2-8 mg of VP-315 administered via intratumor injection into a single target lesion on W1D1. Each 500-μL dose will be divided into 2 injections given at least 15 minutes and no more than 30 minutes apart, with 30% (150 μL) administered in the first injection and the remaining 70% (350 μL) with the second injection. In all parts of the study, the targeted total volume of delivery is 500 μL daily.
  Arms: Part 1 - Cohort 1: Dose Escalation VP-315 2 mg; Part 1 - Cohort 2: Dose Escalation VP-315 3 mg; Part 1 - Cohort 3: Dose Escalation VP-315 4 mg; Part 1 - Cohort 4: Dose Escalation VP-315 5 mg; Part 1 - Cohort 5: Dose Escalation VP-315 6 mg; Part 1 - Cohort 6: Dose Escalation VP-315 7 mg; Part 1 - Cohort 7: Dose Escalation VP-315 8 mg
Drug: Part 2: VP-315 3 Day Dosing/Week - Loading Dose — 4mg (halt the target dose) loading dose on W1D1 administered via intratumor injection into a single target lesion, followed by total daily doses at the full target dose of 8 mg on the remaining days of treatment.
  Arms: Part 2 - Cohort 1: Optimal Dosing Regimen of 3 daily doses of VP-315, 4 mg loading dose
Drug: Part 2: VP-315 3 Day Dosing/Week - No Loading Dose — 8 mg of VP-315 administered daily via intratumor injection into a single target lesion up to 3 consecutive daily doses/week for up to 2 weeks (W1D1, W1D2, W1D3 and W2D1, W2D2, W2D3 - up to 6 total doses).
  Arms: Part 2 - Cohort 2: Optimal Dosing Regimen of 3 daily doses of VP-315 no loading dose
Drug: Part 2: VP-315 2 Day Dosing/Week - Split Dose — 8 mg of VP-315 administered daily via intratumor injection into a single target lesion up to 2 consecutive daily doses/week for up to 2 weeks (W1D1, W1D2, W1D3 and W2D1, W2D2, W2D3 - up to 6 total doses).
  Arms: Part 2 - Cohort 4: Optimal Dosing Regimen of 2 daily doses of VP-315 8 mg (split dose)
Drug: Part 2: VP-315 3 Day Dosing/Week - Split Dose — 8 mg of VP-315 administered daily via intratumor injection into a single target lesion up to 3 consecutive daily doses/week for up to 2 weeks (W1D1, W1D2, W1D3 and W2D1, W2D2, W2D3 - up to 6 total doses).
  Arms: Part 2 - Cohort 5: Optimal Dosing Regimen of 3 daily doses of VP-315 8 mg (split dose)

SUMMARY:
This is a 2-part, open-label, multicenter, dose-escalation, proof-of-concept study with a safety run-in designed to assess the safety, tolerability, MTD, and objective antitumor efficacy of ascending dose strengths of VP-315 when administered intratumorally to adults with biopsy proven basal cell carcinoma (BCC).

The study is expected to enroll approximately 86 subjects with a histological diagnosis of BCC in at least 1 eligible target lesion (confirmed by punch or shave biopsy).

DETAILED DESCRIPTION:
This is a 2-part, open-label, multicenter, dose-escalation, proof-of-concept study with a safety run-in designed to assess the safety, tolerability, maximum tolerated dose (MTD), and objective antitumor efficacy of ascending dose strengths of VP-315 when administered intratumorally to adults with biopsy proven BCC.

The study is expected to enroll approximately 86 subjects with a histological diagnosis of BCC in at least 1 eligible target lesion (confirmed by punch or shave biopsy).

All enrolled subjects will receive VP-315 intradermal injection on an outpatient basis into up to 2 target lesions. In all Parts of the study (1 or 2, as below), each 7-day treatment week comprises up to 3 consecutive treatment days followed by a no-treatment period of at least 4 days. Dosing will commence in a single target lesion. Once a lesion is observed to be fully necrotic (Part 1, Part 2; Cohorts 1-2 only), treatment of that lesion stops, and treatment of subsequent target lesions (up to 2 total) may continue on Day 1 of the following week. In Part 2, Cohorts 4 and 5, treatment of a second target lesion begins on W2D1 (not based on status of necrosis of target lesion 1).

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age
2. Clinically suspected BCC with at least 1 and up to 5 eligible lesion(s) suitable for biopsy and excision
3. Willing to refrain from using nonapproved topical agents on, or within 2 cm of, the target BCC lesions and surrounding areas during the treatment period. Subjects should use topical agents that are gentle (eg, Aquaphor, CeraVe) and will not irritate the skin in these areas.
4. Willing to refrain from exposure to direct sunlight or ultraviolet light and to avoid the use of tanning parlors for the duration of the study
5. Written informed consent obtained, including consent for tissue to be examined by the central dermatopathologist and stored by the Sponsor or designee
6. Willing to undergo BCC surgical excision procedure of target and nontarget BCC lesions after study treatment
7. Willing to delay surgical excision of target and nontarget BCC lesions until the end of treatment (EOT) visit
8. Provides written consent to allow photographs of the target and nontarget BCC lesion to be used as part of the study data
9. Willing to practice a highly effective method of birth control while on study and until 4 weeks after the last treatment. Highly effective birth control includes sexual abstinence, vasectomy, bilateral tubal ligation/occlusion, or a condom with spermicide (men) combined with hormonal birth control or intrauterine device in women.

BCC Lesion Eligibility

Eligible lesions are those that meet the BCC lesion eligibility specifications described herein, from samples that are either from:

* HISTORICAL punch or shave biopsies (i.e., samples collected according to clinical standard of care collected within the 90 days prior to W1D1);
* A 2-mm punch biopsy collected within 90 days of W1D1 for suspected BCC ≥0.5 cm to 1.0 cm, and 3-mm punch biopsy for suspected BCC >1.0 cm to 2.0 cm; or
* A shave biopsy performed according to standard of care to include superficial or middle papillary dermis collected within 90 days of W1D1.

Lesions must meet the following criteria to be eligible for treatment

BCC Lesion Inclusion Criteria

1. For punch biopsies: the size of the lesion(s) must be ≥0.5 cm and </=2 cm in the longest diameter prior to punch biopsy.
2. Histological diagnosis of nodular, micronodular, or superficial BCC, as confirmed by punch or shave biopsy performed within 90 days of W1D1. (NOTE: HISTORICAL punch or shave biopsies are acceptable, provided that the biopsy was performed according to clinical standard of care and was collected within the 90 days prior to Screening.) Subject Exclusion Criteria Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

Exclusion Criteria

1. Presence of known or suspected systemic cancer
2. Treatment with systemic chemotherapeutic agents within the 6 months prior to the screening visit
3. Treatment with systemic immunotherapy, immunomodulators or immunosuppressants within the 12 weeks prior to the screening period
4. Genetic or nevoid conditions (eg, Gorlin / basal cell nevus syndrome, xeroderma pigmentosum)
5. Clinically significant laboratory values, as assessed by the investigator, for the tests listed in the Schedule of Assessments, including:

   1. serum creatinine >1.5× the upper limits of normal and
   2. serum tryptase concentration >11.4 ng/mL
6. Chronic medical condition that in the judgment of the investigator(s) would interfere with the performance of the study or would place the subject at undue risk, such as, but not limited to:

   1. Uncontrolled infection or infection requiring antibiotics
   2. Uncontrolled cardiac failure: Classification III or IV New York Heart Association
   3. Subjects presenting with a systolic BP <110 mmHg and/or diastolic BP <70 mmHg at Screening or Week 1 Day 1 or a history of cerebrovascular or cardiac disorders, or subjects at particular risk of sequelae following a short hypotensive episode.
   4. Uncontrolled systemic or gastrointestinal inflammatory conditions
   5. Known bone marrow dysplasia
   6. History of positive tests for human immunodeficiency virus/acquired immunodeficiency syndrome or active hepatitis B or C
   7. History of systemic autoimmune disease requiring anti-inflammatory or immunosuppressive therapy within 3 months prior to Day 1, with the following exceptions:

   i. Subjects with a history of autoimmune thyroiditis are eligible provided the subject requires only thyroid hormone replacement therapy and disease has been stable for ≥1 year

   ii. Subjects with well-controlled type I diabetes (in the opinion of the investigator) are eligible

   h. Known mast cell activation syndrome, mastocytosis, or chronic idiopathic urticaria
7. Known sensitivity to any of the ingredients in the study medication
8. Elective surgery within 4 weeks prior to the screening visit, during the study, or 4 weeks after the treatment period
9. Evidence of current chronic alcohol or drug abuse
10. Current enrollment in an investigational drug or device study or participation in such a study within 4 weeks of the screening visit
11. In the investigator's opinion, evidence of unwillingness, or inability to follow the restrictions of the protocol and complete the study
12. Females who are pregnant or breastfeeding

BCC Lesion Exclusion Criteria

1. Recurrent or previously treated lesions
2. Lesions within 1 cm of the eyelids or lips, or on the hands, feet, ears, nose, and genitalia
3. Histological evidence of any other tumor in the biopsy specimen
4. Histological evidence of infiltrative, desmoplastic, sclerosing, or morpheaform BCC subtypes in the biopsy specimen
5. Medium- and high-risk basal cell carcinomas as defined by the National Comprehensive Cancer Network (NCCN) or Mohs Appropriate Use Criteria (ie, BCCs eligible for Mohs surgery).

   TARGET LESION EXCLUSION ONLY:
6. For subjects with severe stasis dermatitis, target BCC lesions may not be on the lower extremities
7. Within 2 cm of the target BCC lesion(s):

   1. Treatment with the following topical agents within the 12 weeks prior to the screening visit: aminolevulinic acid, 5-fluorouracil, corticosteroids, diclofenac, imiquimod, ingenol mebutate
   2. Treatment with surgical excision, or curettage within the 2 weeks prior to the screening visit
   3. Evidence of dermatological disease or confounding skin condition that may interfere with clinical evaluation (ie, psoriasis, atopic dermatitis, eczema, propensity to form keloids or hypertrophic scarring)
   4. Use of topical immunomodulators during study
8. Within 5 cm of the target BCC lesion(s): history of any skin cancer, except for other currently identified target and nontarget BCC lesions
9. Target BCC lesion is in the area of prior resurfacing procedure with CO2 laser or any photodynamic and phototherapy treatment within the 3 months prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Bhatia, MD, Principal Investigator — Therapeutics Clinical Research
Locations (13):
- United States (13):
  - Therapeutics Clinical Research, San Diego, California
  - ClearlyDerm, Boca Raton, Florida
  - Life Clinical Trials, Coral Springs, Florida
  - Florida Center for Dermatology, Saint Augustine, Florida
  - Gwinnett Dermatology, Snellville, Georgia
  - Affinity Health, Oakbrook Terrace, Illinois
  - DermAssociates, Rockville, Maryland
  - Lawrence J Green, MD LLC, Rockville, Maryland
  - ActivMed Research - Borthwick, Portsmouth, New Hampshire
  - UPMC St. Margaret, Pittsburgh, Pennsylvania
  - Austin Institute of Clinical Research - Dripping Springs, Dripping Springs, Texas
  - Austin Institute of Clinical Research - Houston, Houston, Texas
  - Austin Institute of Clinical Research - Pflugerville, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Details Study participants were recruited from one of the clinical trial sites selected to participate in the trial that met the study criteria and expressed interest in participating in a BCC trial. Up to 2 Target Lesions for treatment could be enrolled for each participant.
Units Other Than Participants: Target Lesion
Groups:
- Part 1 - Cohort 1 - Intra-subject Dose Escalation: 2 mg VP-315 starting dose. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 2 mg on Day 1, 3 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
- Part 1 - Cohort 2 - Intra-subject Dose Escalation: 3 mg VP-315 starting dose. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 3 mg on Day 1, 4 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
- Part 1 - Cohort 3 - Intra-subject Dose Escalation: 4 mg VP-315 starting dose. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 4 mg on Day 1, 5 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
- Part 1 - Cohort 4 - Intra-subject Dose Escalation: 5 mg VP-315 starting dose. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 5 mg on Day 1, 6 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
- Part 1 - Cohort 5 - Intra-subject Dose Escalation: 6 mg VP-315 starting dose. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 6 mg on Day 1, 7 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
- Part 1 Cohort 6 - Intra-subject Dose Escalation: 7 mg VP-315 starting dose. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 7 mg on Day 1, 8 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
- Part 1 - Cohort 7 - Intra-subject Dose Escalation: 8 mg VP-315 starting dose. Subjects will receive once daily doses of 8 mg for up to 3 days in a 7-day treatment week (e.g., 8 mg on Day 1, 8 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
- Part 2 - Cohort 4 Expansion Optimal Dosing: VP-315 once-daily dosing of 8 mg, administered on 2 consecutive days in one week (W1D1, W1D2). The planned dosing regimen will be a split dose of VP-315 for all treatments. The 500μL (8 mg) dose will be divided into 2 injections given at least 15 minutes and no more than 30 minutes apart, with 30% (150 μL) administered in the first injection and the remaining 70% (350 μL) with the second injection. Treatment for a second Target Lesion may begin on D1 of the next week (W2D1, W2D2). Each individual target lesion is treated for the assigned 2 days only (regardless of necrosis status). Up to 2 target lesions may be treated - up to 4 total doses.
  Part 2: VP-315 2 Day Dosing/Week - Split Dose: 8 mg of VP-315 administered daily via intratumor injection into a single target lesion up to 2 consecutive daily doses/week for up to 2 weeks (W1D1, W1D2, W1D3 and W2D1, W2D2, W2D3 - up to 6 total doses).
- Part 2 - Cohort 5 Expansion: Optimal: VP-315 once-daily dosing of 8 mg, administered on 3 consecutive days in one week (W1D1, W1D2, W1D3). The planned dosing regimen will be a split dose of VP-315 for all treatments. The 500μL (8 mg) dose will be divided into 2 injections given at least 15 minutes and no more than 30 minutes apart, with 30% (150 μL) administered in the first injection and the remaining 70% (350 μL) with the second injection. Treatment for a second target lesion may begin on D1 of the next week (W2D1, W2D2, W2D3). Each individual target lesion is treated for the assigned 3 days only (regardless of necrosis status). Up to 2 target lesions may be treated - up to 6 total doses.
  Part 2: VP-315 3 Day Dosing/Week - Split Dose: 8 mg of VP-315 administered daily via intratumor injection into a single target lesion up to 3 consecutive daily doses/week for up to 2 weeks (W1D1, W1D2, W1D3 and W2D1, W2D2, W2D3 - up to 6 total doses).
Period: Overall Study
Arm/Group | Part 1 - Cohort 1 - Intra-subject Dose Escalation | Part 1 - Cohort 2 - Intra-subject Dose Escalation | Part 1 - Cohort 3 - Intra-subject Dose Escalation | Part 1 - Cohort 4 - Intra-subject Dose Escalation | Part 1 - Cohort 5 - Intra-subject Dose Escalation | Part 1 Cohort 6 - Intra-subject Dose Escalation | Part 1 - Cohort 7 - Intra-subject Dose Escalation | Part 2 - Cohort 1: Optimal Dosing Regimen of 3 Daily Doses of VP-315, 4 mg Loading Dose | Part 2 - Cohort 2: Optimal Dosing Regimen of 3 Daily Doses of VP-315 no Loading Dose | Part 2 - Cohort 4: Optimal Dosing Regimen of 2 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 4 Expansion Optimal Dosing | Part 2 - Cohort 5: Optimal Dosing Regimen of 3 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 5 Expansion: Optimal
Started | 1; 1 Target Lesion | 1; 1 Target Lesion | 1; 1 Target Lesion | 1; 1 Target Lesion (One participant had 2 Target Lesions. Target Lesion 01 was assigned into Cohort 4 and Target Lesion 02 was assigned into Cohort 5. Because of the second lesion, the subject is being counted twice (once in each cohort)) | 1; 1 Target Lesion (One participant had 2 Target Lesions. Target Lesion 01 was assigned into Cohort 4 and Target Lesion 02 was assigned into Cohort 5. Because of the second lesion, the subject is being counted twice (once in each cohort)) | 1; 1 Target Lesion (One participant had 2 Target Lesions. Target Lesion 01 was assigned into Cohort 6 and Target Lesion 02 was assigned into Cohort 7. Because of the second lesion, the subject is being counted twice (once in each cohort)) | 6; 6 Target Lesion (One participant had 2 Target Lesions. Target Lesion 01 was assigned into Cohort 6 and Target Lesion 02 was assigned into Cohort 7. Because of the second lesion, the subject is being counted twice (once in each cohort)) | 6; 7 Target Lesion | 3; 3 Target Lesion | 10; 11 Target Lesion | 26; 31 Target Lesion | 10; 12 Target Lesion | 27; 34 Target Lesion
Completed | 1; 1 Target Lesion | 1; 1 Target Lesion | 1; 1 Target Lesion | 1; 1 Target Lesion (One participant had 2 Target Lesions. Target Lesion 01 was assigned into Cohort 4 and Target Lesion 02 was assigned into Cohort 5. Because of the second lesion, the subject is being counted twice (once in each cohort)) | 1; 1 Target Lesion (One participant had 2 Target Lesions. Target Lesion 01 was assigned into Cohort 4 and Target Lesion 02 was assigned into Cohort 5. Because of the second lesion, the subject is being counted twice (once in each cohort)) | 1; 1 Target Lesion (One participant had 2 Target Lesions. Target Lesion 01 was assigned into Cohort 6 and Target Lesion 02 was assigned into Cohort 7. Because of the second lesion, the subject is being counted twice (once in each cohort)) | 6; 6 Target Lesion (One participant had 2 Target Lesions. Target Lesion 01 was assigned into Cohort 6 and Target Lesion 02 was assigned into Cohort 7. Because of the second lesion, the subject is being counted twice (once in each cohort)) | 6; 7 Target Lesion | 3; 3 Target Lesion | 9; 10 Target Lesion | 25; 30 Target Lesion | 9; 10 Target Lesion | 27; 34 Target Lesion
Not Completed | 0; 0 Target Lesion | 0; 0 Target Lesion | 0; 0 Target Lesion | 0; 0 Target Lesion | 0; 0 Target Lesion | 0; 0 Target Lesion | 0; 0 Target Lesion | 0; 0 Target Lesion | 0; 0 Target Lesion | 1; 1 Target Lesion | 1; 1 Target Lesion | 1; 2 Target Lesion | 0; 0 Target Lesion
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled Subjects. Due to the small number of subjects in each Cohort for Part 1, data are reported with all Part 1 subjects (10) combined per the Statistical Analysis Plan.
Units Other Than Participants: Target Lesions
Groups:
- Part 1 - All Cohorts: Cohorts 1-7: Starting total daily dose of VP-315 was 2-8 mg. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 2 mg on Day 1, 3 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
  Part 1: VP-315 3 Day Dosing/Week: 2-8 mg of VP-315 administered via intratumor injection into a single target lesion on W1D1. Each 500-μL dose will be divided into 2 injections given at least 15 minutes and no more than 30 minutes apart, with 30% (150 μL) administered in the first injection and the remaining 70% (350 μL) with the second injection. In all parts of the study, the targeted total volume of delivery is 500 μL daily.
- Total: Total of all reporting groups
Arm/Group | Part 1 - All Cohorts | Part 2 - Cohort 1: Optimal Dosing Regimen of 3 Daily Doses of VP-315, 4 mg Loading Dose | Part 2 - Cohort 2: Optimal Dosing Regimen of 3 Daily Doses of VP-315 no Loading Dose | Part 2 - Cohort 4: Optimal Dosing Regimen of 2 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 4 Expansion Optimal Dosing | Part 2 - Cohort 5: Optimal Dosing Regimen of 3 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 5 Expansion: Optimal | Total
Number analyzed (Participants) | 10 | 6 | 3 | 10 | 26 | 10 | 27 | 92
Number analyzed (Target Lesions) | 12 | 7 | 3 | 11 | 31 | 12 | 34 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] — Percentage is calculated using the number of subjects in the column heading as the denominator.
  Baseline is defined as the most recent non-missing value prior to study treatment.
  years | 63.4 (7.97) | 63.7 (13.82) | 65.0 (6.08) | 60.4 (10.09) | 66.3 (9.22) | 68.3 (10.59) | 64.2 (9.35) | 64.7 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 1 | 3 | 16 | 5 | 11 | 44
  Male | 5 | 3 | 2 | 7 | 10 | 5 | 16 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 10 | 6 | 3 | 10 | 25 | 10 | 26 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 10 | 6 | 3 | 9 | 26 | 10 | 27 | 91
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 3 | 10 | 26 | 10 | 27 | 92
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Classification of Skin Types I through VI Type I - White skin. Always burns, never tans. Type II - Fair skin. Always burns, tans with difficulty. Type III - Average skin color. Sometimes mild burn, tan about average. Type IV - Light-brown skin. Rarely burns. Tans easily. Type V - Brown skin. Never burns. Tans very easily. Type VI - Black skin. Heavily pigmented. Never burns, tans very easily.
  Participants
    I | 3 | 0 | 0 | 1 | 1 | 3 | 5 | 13
    II | 4 | 6 | 3 | 6 | 20 | 5 | 17 | 61
    III | 3 | 0 | 0 | 3 | 4 | 2 | 5 | 17
    IV | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    V | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    VI | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Target Lesion 01 - Screening Histologic Result [Count of Units; unit: Target Lesions] — Target Lesion 01 - BCC screening histologic result (biopsy pathology result) Population: Data reported for Target Lesion 1
  Target Lesions
    number analyzed (Target Lesions) | 10 | 6 | 3 | 10 | 26 | 10 | 27 | 92
    Micronodular | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Nodular | 4 | 1 | 0 | 4 | 15 | 6 | 15 | 45
    Superficial | 6 | 5 | 3 | 6 | 11 | 4 | 12 | 47
Target Lesion 02 - Screening Histologic Result [Count of Units; unit: Target Lesions] — Population: Target lesion 2 data reported. Number analyzed reflects the participants who had 2 lesions assigned to interventions.
  Target Lesions
    number analyzed (Participants) | 2 | 1 | 0 | 1 | 5 | 2 | 7 | 18
    number analyzed (Target Lesions) | 2 | 1 | 0 | 1 | 5 | 2 | 7 | 18
    Micronodular | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Nodular | 2 | 0 | 0 | 1 | 1 | 1 | 3 | 8
    Superficial | 0 | 1 | 0 | 0 | 4 | 1 | 4 | 10
Target Lesion 01 - Screening BCC Location [Count of Units; unit: Target Lesions] — Population: Target lesion 01 data reported.
  Target Lesions
    number analyzed (Target Lesions) | 10 | 6 | 3 | 10 | 26 | 10 | 27 | 92
    Face or Neck | 1 | 0 | 0 | 1 | 4 | 1 | 4 | 11
    Clavicle or Shoulder | 1 | 0 | 0 | 2 | 5 | 0 | 4 | 12
    Arm | 2 | 1 | 0 | 2 | 7 | 3 | 4 | 19
    Chest or Abdomen | 1 | 0 | 3 | 2 | 5 | 1 | 3 | 15
    Back | 5 | 4 | 0 | 3 | 4 | 3 | 9 | 28
    Buttock or Groin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Leg or Foot | 0 | 1 | 0 | 0 | 1 | 2 | 3 | 7
Target Lesion 02 - Screening BCC Location [Count of Units; unit: Target Lesions] — Population: Target Lesion 02 data reported for participants who had a second lesion assigned to treatment.
  Target Lesions
    number analyzed (Participants) | 2 | 1 | 0 | 1 | 5 | 2 | 7 | 18
    number analyzed (Target Lesions) | 2 | 1 | 0 | 1 | 5 | 2 | 7 | 18
    Face or Neck | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Clavicle or Shoulder | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 5
    Arm | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
    Chest or Abdomen | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 5
    Back | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 4
    Buttocks or Groin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Leg or Foot | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Subjects With Discontinuations Due to Adverse Events
Description: Part 1: Percentage of subjects that discontinued the study due to adverse event
Time Frame: Up to 9 weeks
Population: Part 1 - Enrolled Subjects. Due to the small number of subjects in each Cohort for Part 1, data for Part 1 are reported with all subjects (10) combined per the Statistical Analysis Plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - All Cohorts
Number analyzed (Participants) | 10
Participants | 0

2. Primary Outcome: Part 1: Percentage of Subjects With Dose-limiting Toxicities (DLTs)
Description: Subjects with pre-determined dose-limiting toxicities such as hypotension (specific criteria); significant elevation of serum tryptase; Grade 2 or higher adverse event (with specific criteria)
Time Frame: Day 4 (Safety Assessment)
Population: Safety Population - Part 1 only. Due to the small number of subjects in each Cohort for Part 1, data for Part 1 are reported with all subjects (10) combined per the Statistical Analysis Plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - All Cohorts
Number analyzed (Participants) | 10
Participants | 1

3. Primary Outcome: Part 1: Percentage of Subjects With Cutaneous Reaction by Maximum Severity
Description: Cutaneous injection site reactions are defined as the following preferred terms: Injection site erythema, Injection site induration, Injection site swelling, Injection site vesicles, Injection site exfoliation, Injection site erosion, Injection site ulcer, Injection site necrosis.
  The intended scale for cutaneous injection site reactions is mild, moderate, severe from CRA.
  Subjects having more than one event may appear in more than one System Organ Class or Preferred Term but are counted at most once per each SOC and PT at the maximum severity.
  Cutaneous injection site reactions are types of reactions that can be expected to occur.
Time Frame: Up to 9 weeks
Population: Safety Population. Due to the small number of subjects in each Cohort for Part 1, data for Part 1 are reported with all subjects (10) combined per the Statistical Analysis Plan.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: All Cohorts: Cohorts 1-7: Starting total daily dose of VP-315 was 2-8 mg. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 2 mg on Day 1, 3 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
  Part 1: VP-315 3 Day Dosing/Week: 2-8 mg of VP-315 administered via intratumor injection into a single target lesion on W1D1. Each 500-μL dose will be divided into 2 injections given at least 15 minutes and no more than 30 minutes apart, with 30% (150 μL) administered in the first injection and the remaining 70% (350 μL) with the second injection. In all parts of the study, the targeted total volume of delivery is 500 μL daily.
Arm/Group | Part 1: All Cohorts
Number analyzed (Participants) | 10
Participants
  Erythema: Mild | 1
  Erythema: Moderate | 6
  Erythema: Severe | 0
  Induration: Mild | 4
  Induration: Moderate | 4
  Induration: Severe | 0
  Necrosis: Mild | 0
  Necrosis: Moderate | 4
  Necrosis: Severe | 3
  Swelling: Mild | 4
  Swelling: Moderate | 3
  Swelling: Severe | 0
  Erosion: Mild | 2
  Erosion: Moderate | 4
  Erosion: Severe | 0
  Exfoliation: Mild | 3
  Exfoliation: Moderate | 4
  Exfoliation: Severe | 0
  Ulcer: Mild | 3
  Ulcer: Moderate | 1
  Ulcer: Severe | 1
  Vesicles: Mild | 2
  Vesicles: Moderate | 1
  Vesicles: Severe | 0

4. Primary Outcome: Part 2: Percent of Subjects With Adverse Events
Description: Part 2: Percent of subjects with adverse events, treatment-related AEs
Time Frame: Up to 15 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 - Cohort 1: Optimal Dosing Regimen of 3 Daily Doses of VP-315, 4 mg Loading Dose | Part 2 - Cohort 2: Optimal Dosing Regimen of 3 Daily Doses of VP-315 no Loading Dose | Part 2 - Cohort 4: Optimal Dosing Regimen of 2 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 4 Expansion Optimal Dosing | Part 2 - Cohort 5: Optimal Dosing Regimen of 3 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 5 Expansion: Optimal
Number analyzed (Participants) | 6 | 3 | 10 | 26 | 10 | 27
Participants | 6 | 3 | 10 | 26 | 10 | 25

5. Primary Outcome: Part 2: Percentage of Subjects With Study Discontinuations Due to Adverse Events
Description: Part 2: Percentage of subjects with study discontinuations due to adverse events.
Time Frame: Up to 15 weeks
Population: Enrolled Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 - Cohort 1: Optimal Dosing Regimen of 3 Daily Doses of VP-315, 4 mg Loading Dose | Part 2 - Cohort 2: Optimal Dosing Regimen of 3 Daily Doses of VP-315 no Loading Dose | Part 2 - Cohort 4: Optimal Dosing Regimen of 2 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 4 Expansion Optimal Dosing | Part 2 - Cohort 5: Optimal Dosing Regimen of 3 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 5 Expansion: Optimal
Number analyzed (Participants) | 6 | 3 | 10 | 26 | 10 | 27
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part 2: Percent of Subjects With Treatment Related Adverse Events of Special Interest (TRAEs SI)
Description: Subjects with pre-determined TRAEs of SI such as hypotension (specific criteria); significant elevation of serum tryptase; Grade 2 or higher adverse event (with specific criteria)
Time Frame: Treatment Days up to 2 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 - Cohort 1: Optimal Dosing Regimen of 3 Daily Doses of VP-315, 4 mg Loading Dose | Part 2 - Cohort 2: Optimal Dosing Regimen of 3 Daily Doses of VP-315 no Loading Dose | Part 2 - Cohort 4: Optimal Dosing Regimen of 2 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 4 Expansion Optimal Dosing | Part 2 - Cohort 5: Optimal Dosing Regimen of 3 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 5 Expansion: Optimal
Number analyzed (Participants) | 6 | 3 | 10 | 26 | 10 | 27
Participants
  Hypotension | 0 | 0 | 0 | 1 | 2 | 1
  Blood Pressure Diastolic Decreased | 0 | 0 | 0 | 2 | 0 | 0
  Blood Pressure Systolic Decreased | 0 | 0 | 0 | 1 | 0 | 0
  Injection Site Pain | 1 | 0 | 0 | 0 | 0 | 0
  Injection Site Reaction | 0 | 0 | 0 | 0 | 1 | 0
  Urticaria | 0 | 0 | 0 | 0 | 1 | 0
  Not applicable | 5 | 3 | 10 | 22 | 6 | 26

7. Primary Outcome: Part 2: Percentage of Subjects With Cutaneous Reaction by Maximum Severity
Description: Evaluation of the tissue condition at the treatment site for the presence and severity of each of the following cutaneous reactions; Erythema, Induration, Swelling, Blister Formation, Desquamation, Erosion, Ulceration, Necrosis by a scale of None; Mild; Moderate; Severe. Subjects having more than one event may appear in more than one SOC or PT but are counted at most once per each SOC and PT at the maximum severity.
  Cutaneous injection site reactions are types of reactions that can be expected to occur. The intended scale for cutaneous injection site reactions is mild, moderate, severe from CRA
Time Frame: Up to 105 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 - Cohort 1: Optimal Dosing Regimen of 3 Daily Doses of VP-315, 4 mg Loading Dose | Part 2 - Cohort 2: Optimal Dosing Regimen of 3 Daily Doses of VP-315 no Loading Dose | Part 2 - Cohort 4: Optimal Dosing Regimen of 2 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 4 Expansion Optimal Dosing | Part 2 - Cohort 5: Optimal Dosing Regimen of 3 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 5 Expansion: Optimal
Number analyzed (Participants) | 6 | 3 | 10 | 26 | 10 | 27
Participants
  Erythema: Mild | 5 | 2 | 4 | 13 | 4 | 3
  Erythema: Moderate | 1 | 1 | 6 | 10 | 6 | 19
  Erythema: Severe | 0 | 0 | 0 | 1 | 0 | 4
  Erythema: Not applicable | 0 | 0 | 0 | 2 | 0 | 1
  Induration: Mild | 4 | 1 | 5 | 13 | 6 | 9
  Induration: Moderate | 1 | 0 | 3 | 10 | 3 | 16
  Induration: Severe | 0 | 0 | 0 | 0 | 1 | 1
  Induration: Not applicable | 1 | 2 | 2 | 3 | 0 | 1
  Necrosis: Mild | 0 | 0 | 1 | 5 | 2 | 5
  Necrosis: Moderate | 0 | 2 | 5 | 9 | 7 | 7
  Necrosis: Severe | 4 | 0 | 2 | 5 | 0 | 13
  Necrosis: Not applicable | 2 | 1 | 2 | 7 | 1 | 2
  Swelling: Mild | 3 | 2 | 6 | 7 | 7 | 11
  Swelling: Moderate | 0 | 0 | 3 | 8 | 0 | 13
  Swelling: Severe | 0 | 0 | 0 | 0 | 1 | 0
  Swelling: Not applicable | 3 | 1 | 1 | 11 | 2 | 3
  Erosion: Mild | 1 | 1 | 4 | 3 | 6 | 8
  Erosion: Moderate | 0 | 0 | 0 | 5 | 2 | 6
  Erosion: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Erosion: Not applicable | 5 | 2 | 6 | 18 | 2 | 13
  Exfoliation: Mild | 1 | 1 | 4 | 5 | 3 | 9
  Exfoliation: Moderate | 0 | 0 | 0 | 2 | 1 | 3
  Exfoliation: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Exfoliation: Not applicable | 5 | 2 | 6 | 19 | 6 | 15
  Ulcer: Mild | 1 | 0 | 1 | 4 | 5 | 4
  Ulcer: Moderate | 0 | 0 | 2 | 2 | 3 | 4
  Ulcer: Severe | 0 | 0 | 0 | 0 | 0 | 1
  Ulcer: Not applicable | 5 | 3 | 7 | 20 | 2 | 18
  Vesicles: Mild | 0 | 0 | 1 | 2 | 0 | 3
  Vesicles: Moderate | 0 | 0 | 2 | 0 | 0 | 4
  Vesicles: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Vesicles: Not applicable | 6 | 3 | 7 | 24 | 10 | 20

8. Secondary Outcome: Part 2: Percentage of Subjects With Clinical Clearance of Treated Lesion(s) at Excision
Description: Clinical clearance of Target Lesion at excision as determined by visual assessment (no residual tumor seen on visual inspection). Clinical assessment using Physician Global Assessment (PGA). PGA scale: 100% Improvement, no visible tumor; 75% to less than 100% improvement, 50% to less than 75% improvement, 25% to less than 50% improvement, Up to 25% improvement, No change, Worse.
Time Frame: Day 84-91
Population: Full Analysis Population. Participants with the Physician Global Assessment completed at the End of Treatment Visit. Report is based on Target Lesion 01 and Target Lesion 2 data in separate rows.
Measure: Count of Units; unit: Target Lesions
Units Other Than Participants: Target Lesions
Arm/Group | Part 2 - Cohort 1: Optimal Dosing Regimen of 3 Daily Doses of VP-315, 4 mg Loading Dose | Part 2 - Cohort 2: Optimal Dosing Regimen of 3 Daily Doses of VP-315 no Loading Dose | Part 2 - Cohort 4: Optimal Dosing Regimen of 2 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 4 Expansion Optimal Dosing | Part 2 - Cohort 5: Optimal Dosing Regimen of 3 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 5 Expansion: Optimal
Number analyzed (Participants) | 6 | 3 | 9 | 25 | 9 | 25
Number analyzed (Target Lesions) | 7 | 3 | 9 | 30 | 11 | 31
Target Lesions
  Target Lesion 1: number analyzed (Target Lesions) | 6 | 3 | 9 | 25 | 9 | 25
  Target Lesion 1: 100% Improvement, no visible tumor | 5 | 1 | 6 | 14 | 5 | 19
  Target Lesion 1: 75% to less than 100% improvement | 0 | 1 | 3 | 2 | 2 | 4
  Target Lesion 1: 50% to less than 75% improvement | 0 | 0 | 0 | 4 | 0 | 0
  Target Lesion 1: 25% to less than 50% improvement | 0 | 0 | 0 | 0 | 2 | 0
  Target Lesion 1: Up to 25% improvement | 0 | 0 | 0 | 2 | 0 | 1
  Target Lesion 1: No change | 1 | 1 | 0 | 3 | 0 | 1
  Target Lesion 1: Worse | 0 | 0 | 0 | 0 | 0 | 0
  Target Lesion 2: number analyzed (Participants) | 1 | 0 | 0 | 5 | 2 | 6
  Target Lesion 2: number analyzed (Target Lesions) | 1 | 0 | 0 | 5 | 2 | 6
  Target Lesion 2: 100% Improvement, no visible tumor | 1 | 0 | 0 | 4 | 1 | 5
  Target Lesion 2: 75% to less than 100% improvement | 0 | 0 | 0 | 0 | 0 | 0
  Target Lesion 2: 50% to less than 75% improvement | 0 | 0 | 0 | 0 | 1 | 0
  Target Lesion 2: 25% to less than 50% improvement | 0 | 0 | 0 | 0 | 0 | 0
  Target Lesion 2: Up to 25% improvement | 0 | 0 | 0 | 0 | 0 | 0
  Target Lesion 2: No change | 0 | 0 | 0 | 1 | 0 | 1
  Target Lesion 2: Worse | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Part 2: Percentage of Subjects With Histological Clearance of Treated Lesion(s) at Excision
Description: Percentage of Subjects with histological clearance of treated lesion(s) at excision. Histologic clearance confirmed by central dermatopathologist.
  Percentage is calculated using the number of subjects with non-missing responses within lesion as the denominator.
  *Scar indicates complete histologic clearance
Time Frame: Day 84-91
Population: Full Analysis Population. Participants with Target Lesion(s) excised and histology confirmed by central dermatopathologist. Report is based on Target Lesion 01 and Target Lesion 2 data presented in separate rows. NOTE: All participants had a Target Lesion 1, however, not all participants had a Target Lesion 2, therefore, the numbers are not the same.
Measure: Count of Units; unit: Target Lesions
Units Other Than Participants: Target Lesions
Arm/Group | Part 2 - Cohort 1: Optimal Dosing Regimen of 3 Daily Doses of VP-315, 4 mg Loading Dose | Part 2 - Cohort 2: Optimal Dosing Regimen of 3 Daily Doses of VP-315 no Loading Dose | Part 2 - Cohort 4: Optimal Dosing Regimen of 2 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 4 Expansion Optimal Dosing | Part 2 - Cohort 5: Optimal Dosing Regimen of 3 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 5 Expansion: Optimal
Number analyzed (Participants) | 6 | 3 | 9 | 25 | 9 | 25
Number analyzed (Target Lesions) | 7 | 3 | 9 | 29 | 11 | 31
Target Lesions
  Target Lesion 1: number analyzed (Target Lesions) | 6 | 3 | 9 | 25 | 9 | 25
  Target Lesion 1: Focal Nodular | 0 | 0 | 0 | 0 | 0 | 0
  Target Lesion 1: Micronodular | 0 | 0 | 0 | 0 | 0 | 0
  Target Lesion 1: Nodular | 0 | 1 | 2 | 8 | 1 | 7
  Target Lesion 1: Superficial | 1 | 0 | 0 | 2 | 1 | 1
  Target Lesion 1: Superficial Nodular | 0 | 1 | 2 | 2 | 4 | 3
  Target Lesion 1: Scar (Complete histologic clearance) | 5 | 1 | 5 | 13 | 3 | 14
  Target Lesion 2: number analyzed (Participants) | 1 | 0 | 0 | 4 | 2 | 6
  Target Lesion 2: number analyzed (Target Lesions) | 1 | 0 | 0 | 4 | 2 | 6
  Target Lesion 2: Focal Nodular | 0 | 0 | 0 | 0 | 0 | 0
  Target Lesion 2: Micronodular | 0 | 0 | 0 | 0 | 0 | 0
  Target Lesion 2: Nodular | 0 | 0 | 0 | 1 | 0 | 2
  Target Lesion 2: Superficial | 0 | 0 | 0 | 1 | 0 | 0
  Target Lesion 2: Superficial Nodular | 1 | 0 | 0 | 0 | 1 | 1
  Target Lesion 2: Scar (Complete histologic clearance) | 0 | 0 | 0 | 2 | 1 | 3

10. Secondary Outcome: Part 2: Mean Estimated Remaining Tumor Volume at Excision
Description: Estimate of remaining tumor volume (necrotic cells:tumor cells) at excision by central dermatopathologist
  Scale: 0 = None Remaining to 100 = All Remaining.
Time Frame: Day 84-91
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 2 - Cohort 1: Optimal Dosing Regimen of 3 Daily Doses of VP-315, 4 mg Loading Dose | Part 2 - Cohort 2: Optimal Dosing Regimen of 3 Daily Doses of VP-315 no Loading Dose | Part 2 - Cohort 4: Optimal Dosing Regimen of 2 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 4 Expansion Optimal Dosing | Part 2 - Cohort 5: Optimal Dosing Regimen of 3 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 5 Expansion: Optimal
Number analyzed (Participants) | 6 | 3 | 9 | 25 | 9 | 25
units on a scale
  Target Lesion 1 | 1.7 (4.08) | 11.7 (12.58) | 11.1 (19.49) | 14.8 (22.10) | 22.6 (25.45) | 14.3 (21.00)
  Target Lesion 2: number analyzed (Participants) | 1 | 0 | 0 | 4 | 2 | 6
  Target Lesion 2 | 5.0 |  |  | 6.3 (9.46) | 7.5 (10.61) | 13.3 (27.87)

11. Secondary Outcome: Part 2 (Cohorts 4 and 5 Expansion Groups): Plasma Concentrations of VP-315
Description: Pharmacokinetics (PK) of an 8 mg dose of VP-315 administered with the optimal dosing regimen
Time Frame: Day 1-2
Population: PK Population - Part 2, Cohorts 4 Expansion and 5 Expansion subjects that consented to participate. Includes subjects in Safety Population with quantifiable PK concentration data.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2 - Cohort 4 Expansion Optimal Dosing | Part 2 - Cohort 5 Expansion: Optimal
Number analyzed (Participants) | 9 | 14
h*ng/mL | 32.1 (2.95) | 29.4 (13.78)

ADVERSE EVENTS:
Time Frame: 4-5 months After the informed consent is signed through the end of study follow-up visit. (up to 42 days Screening; treatment in 1-week intervals; surgical excision of all target and nontarget lesions 4 to 6 weeks (Part 1) and 12 to 14 weeks after W1D1 injection; follow-up (F/U) visit at 1- or 2-weeks post excision).
Description: Due to the small number of subjects in each Cohort for Part 1, adverse events for Part 1 are reported with all subjects (10) combined per the Statistical Analysis Plan.
Groups:
- Part 1 - All Cohorts: Due to the small number of subjects in each Cohort for Part 1, adverse events for Part 1 are reported with all subjects (10) combined per the Statistical Analysis Plan. Cohorts 1-7: Starting total daily dose of VP-315 was 2-8 mg. Subjects will receive ascending once daily doses increasing in 1 mg increments for up to 3 days in a 7-day treatment week (e.g., 2 mg on Day 1, 3 mg on Day 2) until the first lesion is necrosed or a DLT occurs. Subjects may be treated for a maximum of 2 weeks and a maximum total daily dose of 8 mg.
  Part 1: VP-315 3 Day Dosing/Week: 2-8 mg of VP-315 administered via intratumor injection into a single target lesion on W1D1. Each 500-μL dose will be divided into 2 injections given at least 15 minutes and no more than 30 minutes apart, with 30% (150 μL) administered in the first injection and the remaining 70% (350 μL) with the second injection. In all parts of the study, the targeted total volume of delivery is 500 μL daily.
Arm/Group | Part 1 - All Cohorts | Part 2 - Cohort 1: Optimal Dosing Regimen of 3 Daily Doses of VP-315, 4 mg Loading Dose | Part 2 - Cohort 2: Optimal Dosing Regimen of 3 Daily Doses of VP-315 no Loading Dose | Part 2 - Cohort 4: Optimal Dosing Regimen of 2 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 4 Expansion Optimal Dosing | Part 2 - Cohort 5: Optimal Dosing Regimen of 3 Daily Doses of VP-315 8 mg (Split Dose) | Part 2 - Cohort 5 Expansion: Optimal
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/3 | 0/10 | 0/26 | 0/10 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/3 | 1/10 | 0/26 | 0/10 | 0/27
Other Adverse Events (participants affected / at risk) | 10/10 | 6/6 | 3/3 | 10/10 | 26/26 | 10/10 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - All Cohorts (N=10) | Part 2 - Cohort 1: Optimal Dosing Regimen of 3 Daily Doses of VP-315, 4 mg Loading Dose (N=6) | Part 2 - Cohort 2: Optimal Dosing Regimen of 3 Daily Doses of VP-315 no Loading Dose (N=3) | Part 2 - Cohort 4: Optimal Dosing Regimen of 2 Daily Doses of VP-315 8 mg (Split Dose) (N=10) | Part 2 - Cohort 4 Expansion Optimal Dosing (N=26) | Part 2 - Cohort 5: Optimal Dosing Regimen of 3 Daily Doses of VP-315 8 mg (Split Dose) (N=10) | Part 2 - Cohort 5 Expansion: Optimal (N=27)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - All Cohorts (N=10) | Part 2 - Cohort 1: Optimal Dosing Regimen of 3 Daily Doses of VP-315, 4 mg Loading Dose (N=6) | Part 2 - Cohort 2: Optimal Dosing Regimen of 3 Daily Doses of VP-315 no Loading Dose (N=3) | Part 2 - Cohort 4: Optimal Dosing Regimen of 2 Daily Doses of VP-315 8 mg (Split Dose) (N=10) | Part 2 - Cohort 4 Expansion Optimal Dosing (N=26) | Part 2 - Cohort 5: Optimal Dosing Regimen of 3 Daily Doses of VP-315 8 mg (Split Dose) (N=10) | Part 2 - Cohort 5 Expansion: Optimal (N=27)
Injection site erythema (General disorders) | 7 (7) | 6 (6) | 3 (3) | 10 (10) | 24 (24) | 10 (10) | 26 (26) — and administration site conditions
Injection site induration (General disorders) | 8 (8) | 5 (5) | 1 (1) | 8 (8) | 23 (23) | 10 (10) | 26 (26) — General disorders and administration site conditions
Injection site necrosis (General disorders) | 7 (7) | 4 (4) | 2 (2) | 8 (8) | 19 (19) | 9 (9) | 25 (25) — General disorders and administration site conditions
Injection site swelling (General disorders) | 7 (7) | 3 (3) | 2 (2) | 8 (8) | 15 (15) | 8 (8) | 24 (24) — General disorders and administration site conditions
Injection site erosion (General disorders) | 6 (6) | 1 (1) | 1 (1) | 4 (4) | 8 (8) | 8 (8) | 14 (14) — General disorders and administration site conditions
Injection site exfoliation (General disorders) | 7 (7) | 1 (1) | 1 (1) | 4 (4) | 7 (7) | 4 (4) | 12 (12) — General disorders and administration site conditions
Injection site ulcer (General disorders) | 5 (5) | 1 (1) | 0 (0) | 3 (3) | 6 (6) | 8 (8) | 9 (9) — General disorders and administration site conditions
Injection site pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 6 (6) | 1 (1) | 8 (8) — General disorders and administration site conditions
Injection site vesicles (General disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 7 (7) — General disorders and administration site conditions
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — General disorders and administration site conditions
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypertrophic Scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Non-small cell lung carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema; Injection site erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — General disorders and administration site conditions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution is restricted from disclosing all data or results which are the sole property of the sponsor and considered confidential information. The Institution may not present data or results without prior Sponsor review and written consent

DOCUMENTS (2):
  • Study Protocol (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT05188729/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT05188729/SAP_001.pdf